CLINICAL TRIAL: NCT00918580
Title: A Phase 3, Open-Label, Single-Arm Trial Evaluating the Safety, Tolerability, and Immunogenicity of 13-valent Pneumococcal Conjugate Vaccine in Children With Sickle Cell Disease Previously Immunized With 23vPS Vaccine
Brief Title: Study Evaluating 13-valent Pneumococcal Conjugate Vaccine (13vPnC) in Children With Sickle Cell Disease
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: 6096A1-3014; B1851013
Record Dates: First submitted 2009-06-09; First posted 2009-06-11 (Estimated); Results first posted 2014-04-21 (Estimated); Last update posted 2014-04-21 (Estimated); Status verified 2014-03

CONDITIONS: Pneumococcal Conjugate Vaccine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- 1 (Experimental)
  Interventions: Biological: 13-valent Pneumoccocal Conjugate Vaccine

INTERVENTIONS:
Biological: 13-valent Pneumoccocal Conjugate Vaccine — 2 doses of 13vPnC will be administered by intramuscular injection separated by approximately 6 months.
  Other Names: 13vPnC

SUMMARY:
This study is to evaluate the safety, tolerability and immunogenicity of 13-valent pneumococcal Conjugate Vaccine in children with Sickle Cell Disease who have already been vaccinated with 23-valent polysaccharide vaccine. The study will measure the amount of antibodies (the proteins that fight off germs) produced by children with Sickle Cell Disease after they have been given the 13-valent pneumococcal vaccine between 6 and less than 18 years of age. They will be given the vaccination twice, each vaccination separated by approximately 6 months.

ELIGIBILITY:
Inclusion Criteria:

* Male or female subject between the ages of >=6 to <18 years.
* Diagnosis of SCD
* 23vPS vaccination at least 6 months prior to enrollment.

Exclusion Criteria:

* Previous vaccination with pneumococcal conjugate vaccine.
* Previous reaction to any vaccine or vaccine-related component or contraindication to vaccination with pneumococcal conjugate vaccine.

Ages: 6 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 158 (Actual)
Dates: Start 2009-11; Primary Completion 2013-03 (Actual); Study Completion 2013-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (14):
- United States (4):
  - Pfizer Investigational Site, Birmingham, Alabama
  - Pfizer Investigational Site, Louisville, Kentucky
  - Pfizer Investigational Site, The Bronx, New York
  - Pfizer Investigational Site, Nashville, Tennessee
- Pfizer Investigational Site, Cairo, Cairo Governorate, Egypt
- Pfizer Investigational Site, Paris, France
- Italy (2):
  - Pfizer Investigational Site, Orbassano (TO)
  - Pfizer Investigational Site, Roma
- Lebanon (2):
  - Pfizer Investigational Site, Beirut, Lebanon
  - Pfizer Investigational Site, Beirut
- Pfizer Investigational Site, Riyadh, Saudi, Saudi Arabia
- United Kingdom (3):
  - Pfizer Investigational Site, Manchester, Cheshire
  - Pfizer Investigational Site, London, United Kingdom
  - Pfizer Investigational Site, London

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=6096A1-3014&StudyName=Study%20Evaluating%2013-valent%20Pneumococcal%20Conjugate%20Vaccine%20%2813vPnC%29%20in%20Children%20with%20Sickle%20Cell%20Disease

RESULTS

PARTICIPANT FLOW:
Groups:
- 13vPnC: Participants previously immunized with 23-valent pneumococcal polysaccharide vaccine (23vPS) received 2 single 0.5 milliliter (mL) doses of 13-valent pneumococcal conjugate vaccine (13vPnC) intramuscular injection, 6 months apart.
Period: Up to 6-month Follow-up(FU)
Arm/Group | 13vPnC
Started | 158
Vaccinated Dose 1 | 158
Vaccinated Dose 2 | 146
Completed | 147 (Completed include 1 participant:withdrew before Dose 2 (protocol violation) but completed 6-month FU)
Not Completed | 11
Not completed — Adverse Event | 1
Not completed — Lost to Follow-up | 5
Not completed — Withdrawal by Subject | 2
Not completed — Parent/Legal Guardian Request | 2
Not completed — Failed to Return | 1
Period: After 6-month FU to 1-year FU
Arm/Group | 13vPnC
Started | 147
Continued After 6-Month FU | 89
Completed | 87
Not Completed | 60
Not completed — Did Not Continue After 6-Month FU | 58
Not completed — Failed to Return | 2

BASELINE CHARACTERISTICS:
Population: All-available immunogenicity (AAI) population included all participants who had at least 1 valid and determinate pneumococcal assay result for the planned analysis.
Arm/Group | 13vPnC
Number analyzed (Participants) | 158
Age, Continuous [Mean (Standard Deviation); unit: years] | 13.3 (3.08)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 76
  Male | 82

OUTCOME MEASURES:

1. Primary Outcome: Geometric Mean Fold Rise (GMFR) in Serotype-Specific Pneumococcal Immunoglobulin G (IgG) From 1 Month After 13vPnC Dose 1 to 1 Month After 13vPnC Dose 2
Description: GMFR for the 13 pneumococcal serotypes (1, 3, 4, 5, 6A, 6B, 7F, 9V, 14, 18C, 19A, 19F, and 23F) from 1 month after 13vPnC Dose 1 to 1 month after 13vPnC Dose 2 were computed using the logarithmically transformed assay results. Confidence interval (CI) for GMFR were back transformations of a CI based on the Student t distribution for the mean logarithm of the mean fold rise. GMFRs were calculated using all participants with available data from both 1 month after 13vPnC Dose 1 and after 13vPnC Dose 2 blood draws. Here number of participants analyzed signifies the evaluable immunogenicity population and "N" signifies participants with a determinate IgG antibody concentration for the given serotype at both 1 Month After 13vPnC Dose 1 and 1 Month After 13vPnC Dose 2 blood draws. Participants may be represented in more than 1 category.
Time Frame: 1 Month After 13vPnC Dose 1, 1 Month After 13vPnC Dose 2
Population: Evaluable immunogenicity population: eligible participants who received all study vaccinations; had valid and determinate assay result; had blood drawn within pre-specified time-frames; had no major protocol violation (including use of prohibited vaccine/medication, immunoglobulins or chronic systemic corticosteroids).
Measure: Geometric Mean (95% Confidence Interval); unit: fold rise
Arm/Group | 13vPnC
Number analyzed (Participants) | 138
fold rise
  Serotype 4 (N = 137) | 0.75 [0.66 to 0.84]
  Serotype 6B (N = 136) | 0.89 [0.78 to 1.02]
  Serotype 9V (N = 136) | 0.82 [0.75 to 0.91]
  Serotype 14 (N = 137) | 0.75 [0.67 to 0.85]
  Serotype 18C (N = 137) | 0.70 [0.62 to 0.80]
  Serotype 19F (N = 136) | 1.05 [0.91 to 1.20]
  Serotype 23F (N = 135) | 0.91 [0.77 to 1.08]
  Serotype 1 (N = 137) | 0.88 [0.77 to 0.99]
  Serotype 3 (N = 134) | 0.82 [0.75 to 0.90]
  Serotype 5 (N = 136) | 0.90 [0.82 to 0.98]
  Serotype 6A (N = 136) | 0.95 [0.82 to 1.10]
  Serotype 7F (N = 137) | 0.75 [0.67 to 0.85]
  Serotype 19A (N = 137) | 0.83 [0.74 to 0.93]

2. Secondary Outcome: Geometric Mean Fold Rise (GMFR) in Serotype-Specific Pneumococcal Immunoglobulin G (IgG) From Before 13vPnC Dose 1 to 1 Month After 13vPnC Dose 1
Description: GMFR for the 13 pneumococcal serotypes (1, 3, 4, 5, 6A, 6B, 7F, 9V, 14, 18C, 19A, 19F, and 23F) from before 13vPnC Dose 1 to 1 month after 13vPnC Dose 1 were computed using the logarithmically transformed assay results. CI for GMFR were back transformations of a CI based on the Student t distribution for the mean logarithm of the mean fold rise. GMFRs were calculated using all participants with available data from before 13vPnC Dose 1 and 1 month after 13vPnC Dose 1 blood draws. Here number of participants analyzed signifies the evaluable immunogenicity population and "N" signifies participants with determinate IgG antibody concentration for the given serotype at both the before 13vPnC Dose 1 and 1 month after 13vPnC Dose 1 blood draws. Participants may be represented in more than 1 category.
Time Frame: Before 13vPnC Dose 1, 1 month after 13vPnC Dose 1
Population: as for outcome 1
Measure: Geometric Mean (95% Confidence Interval); unit: fold rise
Arm/Group | 13vPnC
Number analyzed (Participants) | 138
fold rise
  Serotype 4 (N = 136) | 6.91 [5.27 to 9.06]
  Serotype 6B (N = 137) | 4.72 [3.80 to 5.85]
  Serotype 9V (N = 138) | 3.10 [2.60 to 3.70]
  Serotype 14 (N = 138) | 5.50 [4.05 to 7.46]
  Serotype 18C (N = 137) | 5.58 [4.47 to 6.97]
  Serotype 19F (N = 134) | 4.76 [3.77 to 6.03]
  Serotype 23F (N = 137) | 6.58 [5.12 to 8.46]
  Serotype 1 (N = 129) | 3.60 [2.90 to 4.46]
  Serotype 3 (N = 133) | 2.03 [1.78 to 2.31]
  Serotype 5 (N = 138) | 1.74 [1.56 to 1.94]
  Serotype 6A (N = 132) | 4.10 [3.32 to 5.05]
  Serotype 7F (N = 137) | 4.38 [3.62 to 5.30]
  Serotype 19A (N = 138) | 3.28 [2.73 to 3.96]

3. Secondary Outcome: Geometric Mean Fold Rise (GMFR) in Serotype-Specific Pneumococcal Immunoglobulin G (IgG) From Before 13vPnC Dose 2 to 1 Month After 13vPnC Dose 2
Description: GMFR for the 13 pneumococcal serotypes (1, 3, 4, 5, 6A, 6B, 7F, 9V, 14, 18C, 19A, 19F, and 23F) from before 13vPnC Dose 2 to 1 month after 13vPnC Dose 2 were computed using the logarithmically transformed assay results. CI for GMFR were back transformations of a CI based on the Student t distribution for the mean logarithm of the mean fold rise. GMFRs were calculated using all participants with available data from before 13vPnC Dose 2 and 1 month after 13vPnC Dose 2 blood draws. Here number of participants analyzed signifies the evaluable immunogenicity population and "N" signifies participants with determinate IgG antibody concentration for the given serotype at both the before 13vPnC Dose 2 and 1 month after 13vPnC Dose 2 blood draws. Participants may be represented in more than 1 category.
Time Frame: Before 13vPnC Dose 2, 1 month after 13vPnC Dose 2
Population: as for outcome 1
Measure: Geometric Mean (95% Confidence Interval); unit: fold rise
Arm/Group | 13vPnC
Number analyzed (Participants) | 138
fold rise
  Serotype 4 (N = 137) | 1.86 [1.69 to 2.04]
  Serotype 6B (N = 137) | 1.80 [1.60 to 2.03]
  Serotype 9V (N = 136) | 1.48 [1.37 to 1.59]
  Serotype 14 (N = 137) | 1.24 [1.15 to 1.35]
  Serotype 18C (N = 137) | 1.47 [1.34 to 1.62]
  Serotype 19F (N = 135) | 2.08 [1.85 to 2.34]
  Serotype 23F (N = 135) | 2.04 [1.75 to 2.37]
  Serotype 1 (N = 136) | 1.73 [1.57 to 1.92]
  Serotype 3 (N = 133) | 1.36 [1.25 to 1.47]
  Serotype 5 (N = 135) | 1.30 [1.22 to 1.39]
  Serotype 6A (N = 133) | 1.80 [1.60 to 2.02]
  Serotype 7F (N = 137) | 1.75 [1.61 to 1.90]
  Serotype 19A (N = 137) | 1.48 [1.36 to 1.61]

4. Secondary Outcome: Ratio of Geometric Mean Fold Rise (GMFR) in Serotype-Specific Pneumococcal Immunoglobulin G (IgG) From 13vPnC Dose 1 to 13vPnC Dose 2
Description: GMFR for the 13 pneumococcal serotypes (1, 3, 4, 5, 6A, 6B, 7F, 9V, 14, 18C, 19A, 19F, and 23F) were computed using the logarithmically transformed assay results for Dose 1 (after Dose 1/before Dose 1) and for Dose 2 (after Dose 2/before Dose 2). CI for the ratio of GMFR (Dose 2/Dose 1) were back transformations of a CI based on the Student t distribution for the mean logarithm of the measures (Dose 2 - Dose 1). Here number of participants analyzed signifies the evaluable immunogenicity population and "N" signifies participants with determinate IgG antibody concentration for given serotype at before 13vPnC Dose 1, 1 month after 13vPnC Dose 1, before 13vPnC Dose 2 and 1 month after 13vPnC Dose 2 blood draws. Participants may be represented in more than 1 category.
Time Frame: Before 13vPnC Dose 1, 1 month after 13vPnC Dose 1, before 13vPnC Dose 2, 1 month after 13vPnC Dose 2
Population: as for outcome 1
Measure: Geometric Mean (95% Confidence Interval); unit: ratio of GMFR
Arm/Group | 13vPnC
Number analyzed (Participants) | 138
ratio of GMFR
  Serotype 4 (N = 135) | 0.26 [0.20 to 0.35]
  Serotype 6B (N = 136) | 0.38 [0.29 to 0.49]
  Serotype 9V (N = 136) | 0.49 [0.41 to 0.59]
  Serotype 14 (N = 137) | 0.22 [0.16 to 0.31]
  Serotype 18C (N = 136) | 0.26 [0.21 to 0.34]
  Serotype 19F (N = 132) | 0.44 [0.34 to 0.57]
  Serotype 23F (N = 135) | 0.32 [0.24 to 0.43]
  Serotype 1 (N = 127) | 0.47 [0.37 to 0.59]
  Serotype 3 (N = 130) | 0.66 [0.58 to 0.75]
  Serotype 5 (N = 135) | 0.75 [0.66 to 0.85]
  Serotype 6A (N = 127) | 0.45 [0.35 to 0.58]
  Serotype 7F (N = 136) | 0.39 [0.32 to 0.49]
  Serotype 19A (N = 137) | 0.45 [0.36 to 0.55]

5. Secondary Outcome: Geometric Mean Concentration (GMC) for Serotype-Specific Pneumococcal Immunoglobulin G (IgG) Antibody
Description: Antibody GMC for the 13 pneumococcal serotypes (1, 3, 4, 5, 6A, 6B, 7F, 9V, 14, 18C, 19A, 19F, and 23F) are presented. GMC (13vPnC) and corresponding 2-sided 95 percent (%) CIs were evaluated. Geometric means were calculated using all participants with available data for the specified blood draw. CI for GMC were back transformations of a CI based on the Student t distribution for the mean logarithm of the concentrations. Here number of participants analyzed signifies the evaluable immunogenicity population and "N" signifies participants with determinate IgG antibody concentration for the given serotype at specified time point. Participants may be represented in more than 1 category.
Time Frame: Before 13vPnC Dose 1, 1 month after 13vPnC Dose 1, before 13vPnC Dose 2, 1 month after 13vPnC Dose 2
Population: as for outcome 1
Measure: Geometric Mean (95% Confidence Interval); unit: microgram per milliliter (mcg/mL)
Arm/Group | 13vPnC
Number analyzed (Participants) | 138
microgram per milliliter (mcg/mL)
  Before 13vPnC Dose 1: Serotype 4 (N = 136) | 1.01 [0.80 to 1.27]
  Before 13vPnC Dose 1: Serotype 6B (N = 138) | 5.79 [4.89 to 6.87]
  Before 13vPnC Dose 1: Serotype 9V (N = 138) | 3.01 [2.56 to 3.53]
  Before 13vPnC Dose 1: Serotype 14 (N = 138) | 6.30 [4.78 to 8.30]
  Before 13vPnC Dose 1: Serotype 18C (N = 137) | 1.40 [1.14 to 1.73]
  Before 13vPnC Dose 1: Serotype 19F (N = 134) | 4.46 [3.60 to 5.53]
  Before 13vPnC Dose 1: Serotype 23F (N = 138) | 2.80 [2.38 to 3.30]
  Before 13vPnC Dose 1: Serotype 1 (N = 129) | 1.57 [1.26 to 1.95]
  Before 13vPnC Dose 1: Serotype 3 (N = 133) | 1.02 [0.83 to 1.25]
  Before 13vPnC Dose 1: Serotype 5 (N = 138) | 4.14 [3.58 to 4.78]
  Before 13vPnC Dose 1: Serotype 6A (N = 132) | 4.62 [3.91 to 5.46]
  Before 13vPnC Dose 1: Serotype 7F (N = 137) | 2.16 [1.80 to 2.59]
  Before 13vPnC Dose 1: Serotype 19A (N = 138) | 8.16 [7.03 to 9.48]
  1 Month After 13vPnC Dose 1: Serotype 4 (N = 138) | 6.85 [5.55 to 8.44]
  1 Month After 13vPnC Dose 1: Serotype 6B (N= 137) | 27.25 [22.09 to 33.61]
  1 Month After 13vPnC Dose 1: Serotype 9V (N= 138) | 9.31 [7.83 to 11.07]
  1 Month After 13vPnC Dose 1: Serotype 14 (N = 138) | 34.63 [27.77 to 43.18]
  1 Month After 13vPnC Dose 1: Serotype 18C (N= 138) | 7.83 [6.42 to 9.54]
  1 Month After 13vPnC Dose 1: Serotype 19F (N= 138) | 20.40 [16.03 to 25.95]
  1 Month After 13vPnC Dose 1: Serotype 23F (N= 137) | 18.25 [14.52 to 22.95]
  1 Month After 13vPnC Dose 1: Serotype 1 (N = 138) | 5.24 [4.30 to 6.39]
  1 Month After 13vPnC Dose 1: Serotype 3 (N = 138) | 2.04 [1.76 to 2.38]
  1 Month After 13vPnC Dose 1: Serotype 5 (N = 138) | 7.19 [6.19 to 8.35]
  1 Month After 13vPnC Dose 1: Serotype 6A (N = 138) | 17.61 [14.16 to 21.91]
  1 Month After 13vPnC Dose 1: Serotype 7F (N = 138) | 9.46 [8.17 to 10.94]
  1 Month After 13vPnC Dose 1: Serotype 19A (N= 138) | 26.82 [22.16 to 32.46]
  Before 13vPnC Dose 2: Serotype 4 (N = 138) | 2.77 [2.29 to 3.35]
  Before 13vPnC Dose 2: Serotype 6B (N = 138) | 13.67 [11.23 to 16.63]
  Before 13vPnC Dose 2: Serotype 9V (N = 138) | 5.19 [4.41 to 6.09]
  Before 13vPnC Dose 2: Serotype 14 (N = 138) | 21.07 [17.29 to 25.67]
  Before 13vPnC Dose 2: Serotype 18C (N = 138) | 3.73 [3.10 to 4.49]
  Before 13vPnC Dose 2: Serotype 19F (N = 137) | 10.34 [8.32 to 12.85]
  Before 13vPnC Dose 2: Serotype 23F (N = 137) | 8.07 [6.63 to 9.83]
  Before 13vPnC Dose 2: Serotype 1 (N = 137) | 2.65 [2.21 to 3.19]
  Before 13vPnC Dose 2: Serotype 3 (N = 135) | 1.27 [1.06 to 1.52]
  Before 13vPnC Dose 2: Serotype 5 (N = 137) | 4.91 [4.26 to 5.66]
  Before 13vPnC Dose 2: Serotype 6A (N = 135) | 9.05 [7.48 to 10.95]
  Before 13vPnC Dose 2: Serotype 7F (N = 138) | 4.09 [3.52 to 4.74]
  Before 13vPnC Dose 2: Serotype 19A (N = 138) | 15.13 [12.73 to 17.98]
  1 Month After 13vPnC Dose 2: Serotype 4 (N = 137) | 5.09 [4.28 to 6.04]
  1 Month After 13vPnC Dose 2: Serotype 6B (N= 137) | 24.52 [20.48 to 29.35]
  1 Month After 13vPnC Dose 2: Serotype 9V (N= 136) | 7.46 [6.46 to 8.61]
  1 Month After 13vPnC Dose 2: Serotype 14 (N = 137) | 26.19 [22.11 to 31.03]
  1 Month After 13vPnC Dose 2: Serotype 18C (N= 137) | 5.44 [4.64 to 6.38]
  1 Month After 13vPnC Dose 2: Serotype 19F (N= 136) | 20.56 [17.15 to 24.63]
  1 Month After 13vPnC Dose 2: Serotype 23F (N= 135) | 16.18 [13.27 to 19.73]
  1 Month After 13vPnC Dose 2: Serotype 1 (N = 137) | 4.51 [3.82 to 5.32]
  1 Month After 13vPnC Dose 2: Serotype 3 (N = 134) | 1.67 [1.42 to 1.97]
  1 Month After 13vPnC Dose 2: Serotype 5 (N = 136) | 6.33 [5.58 to 7.17]
  1 Month After 13vPnC Dose 2: Serotype 6A (N = 136) | 16.37 [13.65 to 19.64]
  1 Month After 13vPnC Dose 2: Serotype 7F (N = 137) | 7.06 [6.20 to 8.04]
  1 Month After 13vPnC Dose 2: Serotype 19A (N= 137) | 22.19 [18.94 to 25.99]

6. Secondary Outcome: Geometric Mean Concentration (GMC) for Serotype-Specific Pneumococcal Immunoglobulin G (IgG) Antibody 1 Year After 13vPnC Dose 2
Description: Antibody GMC for the 13 pneumococcal serotypes (1, 3, 4, 5, 6A, 6B, 7F, 9V, 14, 18C, 19A, 19F, and 23F) are presented. GMC (13vPnC) and corresponding 2-sided 95 percent (%) CIs were evaluated. Geometric means were calculated using all participants with available data for the specified blood draw. CI for GMC were back transformations of a CI based on the Student t distribution for the mean logarithm of the concentrations. Here number of participants analyzed signifies the evaluable immunogenicity population at 1-year follow-up and "N" signifies participants with determinate IgG antibody concentration for the given serotype. Participants may be represented in more than 1 category.
Time Frame: 1 year after 13vPnC Dose 2
Population: Evaluable immunogenicity population at 1-year follow-up: eligible participants who received all study vaccinations; had valid and determinate assay result; had blood drawn within pre-specified time-frames; had no major protocol violation (including use of prohibited vaccine/medication, immunoglobulins or chronic systemic corticosteroids).
Measure: Geometric Mean (95% Confidence Interval); unit: mcg/mL
Arm/Group | 13vPnC
Number analyzed (Participants) | 81
mcg/mL
  Serotype 4 (N = 81) | 1.94 [1.51 to 2.48]
  Serotype 6B (N = 81) | 11.77 [9.43 to 14.71]
  Serotype 9V (N = 81) | 4.50 [3.61 to 5.62]
  Serotype 14 (N = 81) | 15.89 [12.47 to 20.26]
  Serotype 18C (N = 81) | 2.64 [2.03 to 3.42]
  Serotype 19F (N = 81) | 9.87 [7.50 to 13.00]
  Serotype 23F (N = 81) | 7.70 [6.15 to 9.63]
  Serotype 1 (N = 79) | 2.12 [1.65 to 2.71]
  Serotype 3 (N = 67) | 1.01 [0.77 to 1.33]
  Serotype 5 (N = 81) | 4.38 [3.58 to 5.37]
  Serotype 6A (N = 81) | 7.94 [6.45 to 9.77]
  Serotype 7F (N = 81) | 3.47 [2.84 to 4.25]
  Serotype 19A (N = 81) | 13.30 [10.62 to 16.65]

7. Secondary Outcome: Serotype-Specific Pneumococcal Opsonophagocytic Activity (OPA) Geometric Mean Titers (GMT)
Description: Antibody GMTs as measured by OPA assay for 13 pneumococcal serotypes (1, 3, 4, 5, 6A, 6B, 7F, 9V, 14, 18C, 19A, 19F, and 23F). GMT and corresponding 2-sided 95% CIs were evaluated. CIs for the GMTs are back transformations of a confidence interval based on the Student t distribution for the mean logarithm of the titers. GMTs were calculated using all participants with available data for the specified blood draw. Here number of participants analyzed signifies the evaluable immunogenicity population and "N" signifies participants with determinate OPA antibody titer for the given serotype at specified time point. Participants may be represented in more than 1 category.
Time Frame: Before 13vPnC Dose 1, 1 month after 13vPnC Dose 1, before 13vPnC Dose 2, 1 month after 13vPnC Dose 2
Population: as for outcome 1
Measure: Geometric Mean (95% Confidence Interval); unit: titer
Arm/Group | 13vPnC
Number analyzed (Participants) | 138
titer
  Before 13vPnC Dose 1: Serotype 4 (N = 105) | 215 [129.6 to 357.2]
  Before 13vPnC Dose 1: Serotype 6B (N = 105) | 626 [377.5 to 1037.4]
  Before 13vPnC Dose 1: Serotype 9V (N = 109) | 234 [137.6 to 398.7]
  Before 13vPnC Dose 1: Serotype 14 (N = 115) | 628 [425.8 to 925.7]
  Before 13vPnC Dose 1: Serotype 18C (N = 95) | 426 [235.7 to 771.4]
  Before 13vPnC Dose 1: Serotype 19F (N = 96) | 94 [55.0 to 160.7]
  Before 13vPnC Dose 1: Serotype 23F (N = 106) | 34 [21.5 to 54.8]
  Before 13vPnC Dose 1: Serotype 1 (N = 131) | 7 [5.7 to 8.8]
  Before 13vPnC Dose 1: Serotype 3 (N = 107) | 13 [10.1 to 17.5]
  Before 13vPnC Dose 1: Serotype 5 (N = 131) | 10 [7.8 to 13.9]
  Before 13vPnC Dose 1: Serotype 6A (N = 116) | 246 [149.0 to 404.8]
  Before 13vPnC Dose 1: Serotype 7F (N = 120) | 344 [220.5 to 537.9]
  Before 13vPnC Dose 1: Serotype 19A (N = 127) | 137 [100.0 to 187.4]
  1 Month After 13vPnC Dose 1: Serotype 4 (N = 108) | 2670 [2128.1 to 3351.1]
  1 Month After 13vPnC Dose 1: Serotype 6B (N= 116) | 7535 [6320.5 to 8983.5]
  1 Month After 13vPnC Dose 1: Serotype 9V (N= 103) | 2312 [1684.0 to 3172.8]
  1 Month After 13vPnC Dose 1: Serotype 14 (N = 117) | 2288 [1906.6 to 2745.0]
  1 Month After 13vPnC Dose 1: Serotype 18C (N= 103) | 4326 [3250.3 to 5756.8]
  1 Month After 13vPnC Dose 1: Serotype 19F (N = 89) | 1429 [1043.5 to 1957.3]
  1 Month After 13vPnC Dose 1: Serotype 23F (N= 106) | 1607 [1227.4 to 2102.7]
  1 Month After 13vPnC Dose 1: Serotype 1 (N = 123) | 56 [41.0 to 77.4]
  1 Month After 13vPnC Dose 1: Serotype 3 (N = 112) | 115 [93.0 to 142.1]
  1 Month After 13vPnC Dose 1: Serotype 5 (N = 121) | 277 [198.4 to 385.8]
  1 Month After 13vPnC Dose 1: Serotype 6A (N = 117) | 7845 [6581.6 to 9349.9]
  1 Month After 13vPnC Dose 1: Serotype 7F (N = 123) | 3348 [2881.9 to 3888.5]
  1 Month After 13vPnC Dose 1: Serotype 19A (N =118) | 1449 [1164.2 to 1804.3]
  Before 13vPnC Dose 2: Serotype 4 (N = 104) | 1331 [1013.9 to 1748.1]
  Before 13vPnC Dose 2: Serotype 6B (N = 108) | 4174 [3513.0 to 4958.3]
  Before 13vPnC Dose 2: Serotype 9V (N = 99) | 1445 [1051.7 to 1985.5]
  Before 13vPnC Dose 2: Serotype 14 (N = 106) | 1652 [1347.8 to 2024.1]
  Before 13vPnC Dose 2: Serotype 18C (N = 101) | 1928 [1281.1 to 2901.0]
  Before 13vPnC Dose 2: Serotype 19F (N = 92) | 516 [338.8 to 785.5]
  Before 13vPnC Dose 2: Serotype 23F (N = 94) | 897 [619.0 to 1300.4]
  Before 13vPnC Dose 2: Serotype 1 (N = 107) | 23 [17.1 to 32.3]
  Before 13vPnC Dose 2: Serotype 3 (N = 120) | 56 [45.5 to 69.9]
  Before 13vPnC Dose 2: Serotype 5 (N = 107) | 98 [69.2 to 140.2]
  Before 13vPnC Dose 2: Serotype 6A (N = 113) | 4005 [3350.6 to 4786.3]
  Before 13vPnC Dose 2: Serotype 7F (N = 112) | 1791 [1427.0 to 2248.6]
  Before 13vPnC Dose 2: Serotype 19A (N = 108) | 677 [544.4 to 843.1]
  1 Month After 13vPnC Dose 2: Serotype 4 (N = 105) | 3051 [2536.7 to 3670.3]
  1 Month After 13vPnC Dose 2: Serotype 6B (N= 107) | 7601 [6392.6 to 9038.6]
  1 Month After 13vPnC Dose 2: Serotype 9V (N = 96) | 3467 [2784.0 to 4317.6]
  1 Month After 13vPnC Dose 2: Serotype 14 (N = 110) | 2081 [1770.5 to 2446.0]
  1 Month After 13vPnC Dose 2: Serotype 18C (N= 103) | 5271 [4267.8 to 6510.1]
  1 Month After 13vPnC Dose 2: Serotype 19F (N = 89) | 1507 [1139.9 to 1992.2]
  1 Month After 13vPnC Dose 2: Serotype 23F (N= 105) | 2330 [1880.4 to 2887.0]
  1 Month After 13vPnC Dose 2: Serotype 1 (N = 106) | 78 [59.5 to 101.2]
  1 Month After 13vPnC Dose 2: Serotype 3 (N = 109) | 105 [87.2 to 127.2]
  1 Month After 13vPnC Dose 2: Serotype 5 (N = 118) | 273 [213.9 to 349.2]
  1 Month After 13vPnC Dose 2: Serotype 6A (N = 111) | 7633 [6439.6 to 9048.6]
  1 Month After 13vPnC Dose 2: Serotype 7F (N = 114) | 3723 [3276.2 to 4230.1]
  1 Month After 13vPnC Dose 2: Serotype 19A (N= 115) | 1314 [1084.4 to 1592.6]

8. Secondary Outcome: Serotype-Specific Pneumococcal Opsonophagocytic Activity (OPA) Geometric Mean Titers (GMT) 1 Year After 13vPnC Dose 2
Description: Antibody GMTs as measured by OPA assay for 13 pneumococcal serotypes (1, 3, 4, 5, 6A, 6B, 7F, 9V, 14, 18C, 19A, 19F, and 23F). GMT and corresponding 2-sided 95% CIs were evaluated. CIs for the GMTs are back transformations of a confidence interval based on the Student t distribution for the mean logarithm of the titers. GMTs were calculated using all participants with available data for the specified blood draw. Here number of participants analyzed signifies the evaluable immunogenicity population at 1-year follow-up and "N" signifies participants with determinate OPA antibody titer for the given serotype. Participants may be represented in more than 1 category.
Time Frame: 1 year after 13vPnC Dose 2
Population: as for outcome 6
Measure: Geometric Mean (95% Confidence Interval); unit: titer
Arm/Group | 13vPnC
Number analyzed (Participants) | 81
titer
  Serotype 4 (N = 58) | 1107 [764.4 to 1602.2]
  Serotype 6B (N = 59) | 3412 [2746.4 to 4238.7]
  Serotype 9V (N = 66) | 1690 [1157.8 to 2465.5]
  Serotype 14 (N = 64) | 1595 [1281.6 to 1984.9]
  Serotype 18C (N = 59) | 1604 [1107.2 to 2324.2]
  Serotype 19F (N = 55) | 620 [376.6 to 1020.4]
  Serotype 23F (N = 58) | 924 [654.2 to 1306.1]
  Serotype 1 (N = 73) | 25 [17.5 to 35.4]
  Serotype 3 (N = 72) | 31 [22.6 to 42.6]
  Serotype 5 (N = 71) | 102 [70.5 to 148.0]
  Serotype 6A (N = 72) | 2485 [1921.2 to 3214.3]
  Serotype 7F (N = 73) | 2166 [1861.4 to 2519.3]
  Serotype 19A (N = 73) | 589 [449.4 to 771.1]

9. Other Pre Specified Outcome: Percentage of Participants With Prespecified Local Reactions: 13vPnC Dose 1
Description: Specific local reactions were prompted for each day, and reported using an electronic diary. Redness and Swelling were scaled as: Any (redness present or swelling present); Mild (less than <2.5 centimeters [cm] for participants aged 6 to <12 years and 2.5 to 5.0 cm for participants aged greater than or equal to [>=] 12 years); Moderate (2.5 to 7.0 cm for participants aged 6 to <12 years and 5.1 to 10.0 cm for participants aged >=12 years); Severe (>7 cm for participants aged 6 to <12 years and >10 cm for participants aged >=12 years). Pain was scaled as: Any (pain present); Mild (did not interfere with activity); Moderate (interfered with activity); Severe (prevented daily activity). Here "Number of participants analyzed" signifies the safety population for Dose 1 and "N" signifies those participants who reported "Yes" for at least 1 day or "No" for all days for specified local reaction. Participants may be represented in more than 1 category.
Time Frame: Within 7 days after 13vPnC Dose 1
Population: Safety population for Dose 1 included all participants who received Dose 1 of study vaccine and had safety data available.
Measure: Number; unit: percentage of participants
Arm/Group | 13vPnC
Number analyzed (Participants) | 158
percentage of participants
  Pain: Any (N = 144) | 89.6
  Pain: Mild (N = 132) | 81.8
  Pain: Moderate (N = 113) | 56.6
  Pain: Severe (N = 90) | 11.1
  Redness: Any (N = 93) | 23.7
  Redness: Mild (N = 93) | 20.4
  Redness: Moderate (N = 90) | 8.9
  Redness: Severe (N = 87) | 1.1
  Swelling: Any (N = 108) | 49.1
  Swelling: Mild (N = 101) | 37.6
  Swelling: Moderate (N = 100) | 26.0
  Swelling: Severe (N = 87) | 1.1

10. Other Pre Specified Outcome: Percentage of Participants With Prespecified Local Reactions: 13vPnC Dose 2
Description: Specific local reactions were prompted for each day, and reported using an electronic diary. Redness and Swelling were scaled as: Any (redness present or swelling present); Mild (<2.5 cm for participants aged 6 to <12 years and 2.5 to 5.0 cm for participants aged >=12 years); Moderate (2.5 to 7.0 cm for participants aged 6 to <12 years and 5.1 to 10.0 cm for participants aged >=12 years); Severe (>7 cm for participants aged 6 to <12 years and >10 cm for participants aged >=12 years). Pain was scaled as: Any (pain present); Mild (did not interfere with activity); Moderate (interfered with activity); Severe (prevented daily activity). Here number of participants analyzed signifies the safety population for Dose 2 and "N" signifies those participants who reported "Yes" for at least 1 day or "No" for all days for specified local reaction. Participants may be represented in more than 1 category.
Time Frame: Within 7 days after 13vPnC Dose 2
Population: Safety population for Dose 2 included all participants who received Dose 2 of study vaccine and had safety data available.
Measure: Number; unit: percentage of participants
Arm/Group | 13vPnC
Number analyzed (Participants) | 140
percentage of participants
  Pain: Any (N = 111) | 85.6
  Pain: Mild (N = 103) | 77.7
  Pain: Moderate (N = 82) | 53.7
  Pain: Severe (N = 69) | 15.9
  Redness: Any (N = 67) | 26.9
  Redness: Mild (N = 66) | 15.2
  Redness: Moderate (N = 64) | 14.1
  Redness: Severe (N = 63) | 0.0
  Swelling: Any (N = 84) | 53.6
  Swelling: Mild (N = 77) | 37.7
  Swelling: Moderate (N = 73) | 35.6
  Swelling: Severe (N = 63) | 0.0

11. Other Pre Specified Outcome: Percentage of Participants With Prespecified Systemic Events: 13vPnC Dose 1
Description: Specific systemic events (fever >=38 degrees Celsius[C], vomiting, diarrhea, headache, fatigue, muscle pain, joint pain, use of antipyretic medications) were prompted for each day and reported using an electronic diary. Fatigue, headache, muscle pain and joint pain were scaled as: Any(symptom present); Mild(did not interfere with activity); Moderate(some interference); Severe(prevented routine daily activity). Vomiting was scaled as: Any(vomiting present); Mild(1-2 times in 24 hours); Moderate(>2 times in 24 hours); Severe(required intravenous hydration). Diarrhea was scaled as: Any(diarrhea present); Mild(2-3 loose stools in 24 hours);Moderate(4-5 loose stools 24 hours); Severe(>=6 loose stools in 24 hours). Here number of participants analyzed signifies the safety population for Dose 1 and "N" signifies those participants who reported "Yes" for at least 1 day or "No" for all days for specified systemic event. Participants may be represented in more than 1 category.
Time Frame: Within 7 days after 13vPnC Dose 1
Population: as for outcome 9
Measure: Number; unit: percentage of participants
Arm/Group | 13vPnC
Number analyzed (Participants) | 158
percentage of participants
  Fever: >=38, =<38.4 degrees C (N = 81) | 13.6
  Fever: >38.4, =<38.9 degrees C (N = 82) | 7.3
  Fever: >38.9, =<40 degrees C (N = 79) | 3.8
  Fever: >40 degrees C (N = 79) | 1.3
  Vomiting: Any (N = 91) | 15.4
  Vomiting: Mild (N = 89) | 11.2
  Vomiting: Moderate (N = 90) | 6.7
  Vomiting: Severe (N = 87) | 0.0
  Diarrhea: Any (N = 90) | 13.3
  Diarrhea: Mild (N = 87) | 6.9
  Diarrhea: Moderate (N = 90) | 6.7
  Diarrhea: Severe (N = 87) | 2.3
  Headache: Any (N = 110) | 53.6
  Headache: Mild (N = 105) | 42.9
  Headache: Moderate (N = 101) | 34.7
  Headache: Severe (N = 92) | 12.0
  Fatigue: Any (N = 118) | 66.1
  Fatigue: Mild (N = 108) | 48.1
  Fatigue: Moderate (N = 104) | 44.2
  Fatigue: Severe (N = 90) | 14.4
  Muscle Pain: Any (N = 127) | 74.8
  Muscle Pain: Mild (N = 114) | 58.8
  Muscle Pain: Moderate (N = 108) | 47.2
  Muscle Pain: Severe (N = 89) | 10.1
  Joint Pain: Any (N = 103) | 39.8
  Joint Pain: Mild (N = 98) | 23.5
  Joint Pain: Moderate (N = 94) | 23.4
  Joint Pain: Severe (N = 89) | 4.5
  Use of Antipyretic Medications (N = 110) | 58.2

12. Other Pre Specified Outcome: Percentage of Participants With Prespecified Systemic Events: 13vPnC Dose 2
Description: Specific systemic events (fever >=38 degrees C, vomiting, diarrhea, headache, fatigue, muscle pain, joint pain, and use of antipyretic medications) were prompted for each day, and reported using an electronic diary. Fatigue, headache, muscle pain and joint pain were scaled as: Any(symptom present); Mild(did not interfere with activity); Moderate(some interference); Severe(prevented routine daily activity). Vomiting was scaled as: Any(vomiting present); Mild(1-2 times in 24 hours); Moderate(>2 times in 24 hours); Severe (required intravenous hydration). Diarrhea was scaled as: Any(diarrhea present); Mild(2-3 loose stools in 24 hours); Moderate(4-5 loose stools 24 hours); Severe(>=6 loose stools in 24 hours). Here number of participants analyzed signifies the safety population for Dose 2 and "N" signifies those participants who reported "Yes" for at least 1 day or "No" for all days for specified systemic event. Participants may be represented in more than 1 category.
Time Frame: Within 7 days after 13vPnC Dose 2
Population: as for outcome 10
Measure: Number; unit: percentage of participants
Arm/Group | 13vPnC
Number analyzed (Participants) | 140
percentage of participants
  Fever: >=38, =<38.4 degrees C (N = 63) | 9.5
  Fever: >38.4, =<38.9 degrees C (N = 59) | 6.8
  Fever: >38.9, =<40 degrees C (N = 63) | 6.3
  Fever: >40 degrees C (N = 60) | 1.7
  Vomiting: Any (N = 67) | 13.4
  Vomiting: Mild (N = 65) | 9.2
  Vomiting: Moderate (N = 64) | 4.7
  Vomiting: Severe (N = 64) | 1.6
  Diarrhea: Any (N = 68) | 25.0
  Diarrhea: Mild (N = 68) | 19.1
  Diarrhea: Moderate (N = 66) | 12.1
  Diarrhea: Severe (N = 63) | 3.2
  Headache: Any (N = 86) | 59.3
  Headache: Mild (N = 74) | 41.9
  Headache: Moderate (N = 76) | 36.8
  Headache: Severe (N = 66) | 10.6
  Fatigue: Any (N = 96) | 62.5
  Fatigue: Mild (N = 84) | 48.8
  Fatigue: Moderate (N = 83) | 41.0
  Fatigue: Severe (N = 67) | 13.4
  Muscle Pain: Any (N = 98) | 75.5
  Muscle Pain: Mild (N = 87) | 60.9
  Muscle Pain: Moderate (N = 84) | 45.2
  Muscle Pain: Severe (N = 67) | 16.4
  Joint Pain: Any (N = 78) | 44.9
  Joint Pain: Mild (N = 72) | 34.7
  Joint Pain: Moderate (N = 70) | 21.4
  Joint Pain: Severe (N = 65) | 6.2
  Use of Antipyretic Medications (N = 78) | 43.6

ADVERSE EVENTS:
Time Frame: SAEs: 13vPnC Dose 1 through 1-year follow-up after 13vPnC Dose 2. AEs: 13vPnC Dose 1; 13vPnC Dose 2; 6-month follow-up after 13vPnC Dose 2; 1-year follow-up after 13vPnC Dose 2. Local reactions/systemic events: within 7 days after 13vPnC Dose 1 and Dose 2
Description: Safety populations: participants who received at least 1 dose and had safety data available. SAEs and AEs were grouped by system organ class and summarized. AEs included events collected in electronic diary (local and systemic reactions; systematic assessment) and events collected on case report form at each visit (nonsystematic assessment).
Groups:
- 13vPnC Dose 1: Participants previously immunized with 23vPS who received a single 0.5 mL dose of 13vPnC intramuscular injection on Day 1 (13vPnC Dose 1), assessed between 13vPnC Dose 1 and before 13vPnC Dose2.
- 13vPnC Dose 2: Participants previously immunized with 23vPS who received Dose 2 of 0.5 mL 13vPnC intramuscular injection, assessed between 13vPnC Dose 2 and before 13vPnC Dose 2 blood draw.
- 6-Month Follow-up: Participants previously immunized with 23vPS who received at least 1 of the 2 single 0.5 mL doses of 13vPnC intramuscular injection, 6 months apart, assessed from last 13vPnC Dose (Dose 1 or Dose 2) blood draw to the 6-month follow-up telephone contact.
- 1-Year Follow-up: Participants previously immunized with 23vPS who received 2 single 0.5 mL doses of 13vPnC intramuscular injection, 6 months apart, assessed from the 6-month follow-up telephone contact after 13vPnC Dose 2 to the 1-year follow-up after 13vPnC Dose 2.
Arm/Group | 13vPnC Dose 1 | 13vPnC Dose 2 | 6-Month Follow-up | 1-Year Follow-up
Serious Adverse Events (participants affected / at risk) | 40/158 | 11/140 | 28/147 | 16/87
Other Adverse Events (participants affected / at risk) | 133/158 | 100/140 | 1/147 | 1/87
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | 13vPnC Dose 1 (N=158) | 13vPnC Dose 2 (N=140) | 6-Month Follow-up (N=147) | 1-Year Follow-up (N=87)
Anaemia (Blood and lymphatic system disorders) | 1 | 0 | 0 | 0
Lymphadenopathy (Blood and lymphatic system disorders) | 1 | 0 | 0 | 0
Haemolytic anaemia (Blood and lymphatic system disorders) | 0 | 0 | 1 | 0
Hypersplenism (Blood and lymphatic system disorders) | 0 | 0 | 1 | 0
Sickle cell anaemia with crisis (Congenital, familial and genetic disorders) | 22 | 5 | 17 | 11
Visual impairment (Eye disorders) | 1 | 0 | 0 | 0
Abdominal pain (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Constipation (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Gastritis (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Gingivitis (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Hiatus hernia (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Nausea (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Oesophagitis (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Pyrexia (General disorders) | 5 | 0 | 2 | 3
Fatigue (General disorders) | 1 | 0 | 0 | 0
Pain (General disorders) | 1 | 0 | 2 | 1
Chest pain (General disorders) | 0 | 0 | 1 | 0
Oedema peripheral (General disorders) | 0 | 0 | 0 | 1
Cholecystitis (Hepatobiliary disorders) | 1 | 0 | 0 | 0
Cholecystitis acute (Hepatobiliary disorders) | 1 | 0 | 0 | 1
Hyperbilirubinaemia (Hepatobiliary disorders) | 1 | 0 | 0 | 0
Upper respiratory tract infection (Infections and infestations) | 2 | 0 | 0 | 0
Bacteraemia (Infections and infestations) | 1 | 0 | 0 | 0
Bronchitis (Infections and infestations) | 1 | 0 | 1 | 1
Device related infection (Infections and infestations) | 1 | 0 | 0 | 0
Osteomyelitis (Infections and infestations) | 1 | 0 | 0 | 1
Pharyngitis (Infections and infestations) | 1 | 0 | 0 | 0
Pharyngotonsillitis (Infections and infestations) | 1 | 0 | 0 | 0
Pneumonia (Infections and infestations) | 1 | 0 | 2 | 4
Pyelonephritis (Infections and infestations) | 1 | 0 | 0 | 0
Tonsillitis (Infections and infestations) | 1 | 0 | 0 | 0
Urinary tract infection (Infections and infestations) | 1 | 0 | 0 | 1
Gastroenteritis (Infections and infestations) | 0 | 0 | 1 | 1
Groin abscess (Infections and infestations) | 0 | 0 | 1 | 0
Hepatitis A (Infections and infestations) | 0 | 0 | 1 | 0
Sinusitis (Infections and infestations) | 0 | 0 | 1 | 0
Staphylococcal bacteraemia (Infections and infestations) | 0 | 0 | 1 | 0
Bone abscess (Infections and infestations) | 0 | 0 | 0 | 1
Rib fracture (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0
Overdose (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0
Hypocalcaemia (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 2 | 0 | 1 | 0
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 | 2 | 0 | 0
Pain in jaw (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 0 | 1 | 1 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0
Flank pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0
Muscular weakness (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0
Headache (Nervous system disorders) | 1 | 0 | 1 | 0
Lethargy (Nervous system disorders) | 1 | 0 | 0 | 0
Migraine (Nervous system disorders) | 1 | 0 | 0 | 0
Cerebral infarction (Nervous system disorders) | 0 | 0 | 1 | 0
Hypoaesthesia (Nervous system disorders) | 0 | 0 | 1 | 0
Unresponsive to stimuli (Nervous system disorders) | 0 | 0 | 1 | 0
Cerebrovascular accident (Nervous system disorders) | 0 | 0 | 0 | 1
Pregnancy (Pregnancy, puerperium and perinatal conditions) | 0 | 2 | 0 | 0
Mental status changes (Psychiatric disorders) | 1 | 0 | 0 | 0
Dysuria (Renal and urinary disorders) | 1 | 0 | 0 | 0
Haematuria (Renal and urinary disorders) | 0 | 0 | 1 | 1
Renal failure (Renal and urinary disorders) | 0 | 0 | 1 | 0
Renal failure chronic (Renal and urinary disorders) | 0 | 0 | 1 | 0
Priapism (Reproductive system and breast disorders) | 1 | 0 | 0 | 0
Acute chest syndrome (Respiratory, thoracic and mediastinal disorders) | 3 | 0 | 2 | 1
Asthma (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 1 | 1
Lung infiltration (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0
Vascular occlusion (Vascular disorders) | 3 | 2 | 0 | 0
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk, or affected / at risk where a term's number at risk differs:
Term (organ system) | 13vPnC Dose 1 (N=158) | 13vPnC Dose 2 (N=140) | 6-Month Follow-up (N=147) | 1-Year Follow-up (N=87)
Sickle cell anaemia with crisis (Congenital, familial and genetic disorders) | 4 | 1 | 0 | 0
Vertigo (Ear and labyrinth disorders) | 0 | 1 | 0 | 0
Conjunctivitis allergic (Eye disorders) | 1 | 0 | 0 | 0
Periorbital oedema (Eye disorders) | 1 | 1 | 0 | 0
Ocular icterus (Eye disorders) | 0 | 1 | 0 | 0
Diarrhoea (Gastrointestinal disorders) | 2 | 0 | 0 | 0
Vomiting (Gastrointestinal disorders) | 2 | 0 | 0 | 0
Abdominal pain upper (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Constipation (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Nausea (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Pancreatic calcification (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Abdominal pain (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Gingival pain (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Oral pain (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Hiatus hernia (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Pyrexia (General disorders) | 5 | 1 | 0 | 0
Chest pain (General disorders) | 2 | 0 | 0 | 0
Injection site pain (General disorders) | 1 | 0 | 0 | 0
Asthenia (General disorders) | 1 | 0 | 0 | 0
Injection site erythema (General disorders) | 1 | 0 | 0 | 0
Injection site movement impairment (General disorders) | 1 | 0 | 0 | 0
Oedema peripheral (General disorders) | 1 | 0 | 0 | 0
Swelling (General disorders) | 1 | 0 | 0 | 0
Injection site swelling (General disorders) | 0 | 1 | 0 | 0
Pain (General disorders) | 0 | 1 | 0 | 0
Cholelithiasis (Hepatobiliary disorders) | 2 | 0 | 0 | 0
Nasopharyngitis (Infections and infestations) | 2 | 0 | 0 | 0
Infection (Infections and infestations) | 1 | 0 | 0 | 0
Pharyngitis (Infections and infestations) | 1 | 1 | 0 | 0
Rhinitis (Infections and infestations) | 1 | 0 | 0 | 0
Viral upper respiratory tract infection (Infections and infestations) | 1 | 0 | 0 | 0
Transfusion reaction (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0
Pain in extremity (Musculoskeletal and connective tissue disorders) | 2 | 2 | 0 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 1 | 1 | 0 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0
Joint swelling (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0
Headache (Nervous system disorders) | 4 | 1 | 0 | 0
Convulsion (Nervous system disorders) | 1 | 0 | 0 | 0
Hypoaesthesia (Nervous system disorders) | 1 | 0 | 0 | 0
Moyamoya disease (Nervous system disorders) | 1 | 0 | 0 | 0
Depression (Psychiatric disorders) | 1 | 0 | 0 | 0
Insomnia (Psychiatric disorders) | 1 | 0 | 0 | 0
Listless (Psychiatric disorders) | 0 | 1 | 0 | 0
Renal failure chronic (Renal and urinary disorders) | 1 | 0 | 0 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 2 | 0 | 0 | 0
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 2 | 0 | 0 | 0
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0
Nasal congestion (Reproductive system and breast disorders) | 1 | 0 | 0 | 0
Productive cough (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0
Rhinitis allergic (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0
Swelling face (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0
Vascular occlusion (Vascular disorders) | 4 | 0 | 0 | 0
Hypertension (Vascular disorders) | 1 | 0 | 0 | 0
Pain (Any) (Skin and subcutaneous tissue disorders) | 129/144 | 95/111 | 0/0 | 0/0
Pain (Mild) (Skin and subcutaneous tissue disorders) | 108/132 | 80/103 | 0/0 | 0/0
Pain (Moderate) (Skin and subcutaneous tissue disorders) | 64/113 | 44/82 | 0/0 | 0/0
Pain (Severe) (Skin and subcutaneous tissue disorders) | 10/90 | 11/69 | 0/0 | 0/0
Redness (Any) (Skin and subcutaneous tissue disorders) | 22/93 | 18/67 | 0/0 | 0/0
Redness (Mild) (Skin and subcutaneous tissue disorders) | 19/93 | 10/66 | 0/0 | 0/0
Redness (Moderate) (Skin and subcutaneous tissue disorders) | 8/90 | 9/64 | 0/0 | 0/0
Redness (Severe) (Skin and subcutaneous tissue disorders) | 1/87 | 0/63 | 0/0 | 0/0
Swelling (Any) (Skin and subcutaneous tissue disorders) | 53/108 | 45/84 | 0/0 | 0/0
Swelling (Mild) (Skin and subcutaneous tissue disorders) | 38/101 | 29/77 | 0/0 | 0/0
Swelling (Moderate) (Skin and subcutaneous tissue disorders) | 26/100 | 26/73 | 0/0 | 0/0
Swelling (Severe) (Skin and subcutaneous tissue disorders) | 1/87 | 0/63 | 0/0 | 0/0
Fever >=38°C but =<38.4°C (General disorders) | 11/81 | 6/63 | 0/0 | 0/0
Fever >38.4°C but =<38.9°C (General disorders) | 6/82 | 4/59 | 0/0 | 0/0
Fever >38.9°C but =<40.0°C (General disorders) | 3/79 | 4/63 | 0/0 | 0/0
Fever >40.0°C (General disorders) | 1/79 | 1/60 | 0/0 | 0/0
Vomiting (Any) (General disorders) | 14/91 | 9/67 | 0/0 | 0/0
Vomiting (Mild) (General disorders) | 10/89 | 6/65 | 0/0 | 0/0
Vomiting (Moderate) (General disorders) | 6/90 | 3/64 | 0/0 | 0/0
Vomiting (Severe) (General disorders) | 0/87 | 1/64 | 0/0 | 0/0
Diarrhea (Any) (General disorders) | 12/90 | 17/68 | 0/0 | 0/0
Diarrhea (Mild) (General disorders) | 6/87 | 13/68 | 0/0 | 0/0
Diarrhea (Moderate) (General disorders) | 6/90 | 8/66 | 0/0 | 0/0
Diarrhea (Severe) (General disorders) | 2/87 | 2/63 | 0/0 | 0/0
Headache (Any) (General disorders) | 59/110 | 51/86 | 0/0 | 0/0
Headache (Mild) (General disorders) | 45/105 | 31/74 | 0/0 | 0/0
Headache (Moderate) (General disorders) | 35/101 | 28/76 | 0/0 | 0/0
Headache (Severe) (General disorders) | 11/92 | 7/66 | 0/0 | 0/0
Fatigue (Any) (General disorders) | 78/118 | 60/96 | 0/0 | 0/0
Fatigue (Mild) (General disorders) | 52/108 | 41/84 | 0/0 | 0/0
Fatigue (Moderate) (General disorders) | 46/104 | 34/83 | 0/0 | 0/0
Fatigue (Severe) (General disorders) | 13/90 | 9/67 | 0/0 | 0/0
Muscle pain (Any) (General disorders) | 95/127 | 74/98 | 0/0 | 0/0
Muscle pain (Mild) (General disorders) | 67/114 | 53/87 | 0/0 | 0/0
Muscle pain (Moderate) (General disorders) | 51/108 | 38/84 | 0/0 | 0/0
Muscle pain (Severe) (General disorders) | 9/89 | 11/67 | 0/0 | 0/0
Joint pain (Any) (General disorders) | 41/103 | 35/78 | 0/0 | 0/0
Joint pain (Mild) (General disorders) | 23/98 | 25/72 | 0/0 | 0/0
Joint pain (Moderate) (General disorders) | 22/94 | 15/70 | 0/0 | 0/0
Joint pain (Severe) (General disorders) | 4/89 | 4/65 | 0/0 | 0/0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Pfizer has the right to review disclosures, requesting a delay of less than 60 days. Investigator will postpone single center publications until after disclosure of pooled data (all sites), less than 12 months from study completion/termination at all participating sites. Investigator may not disclose previously undisclosed confidential information other than study results.